CLINICAL TRIAL: NCT03547934
Title: Safety and Efficacy of Noninvasive Repetitive Pulse Magnetic Stimulation (rPMS) for Fat Disruption of the Abdomen
Brief Title: Fat Reduction Induced by Magnetic Device - Waist Circumference Evaluation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: It wasn't possible to recruit the desired number of patients.
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-Abdomen_004
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Fat Burn
Keywords: Abdominal fat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment Group (Experimental): Treatment with the investigated device - High Intensity Focused ElectroMagnetic System
  Interventions: Device: High Intensity Focused ElectroMagnetic system.

INTERVENTIONS:
Device: High Intensity Focused ElectroMagnetic system. — The treatment administration phase will consist of four (4) treatments, delivered twice a week. The applicator will be applied over the abdomen area. Visible contractions will be induced by the device.

SUMMARY:
The study is a prospective multi-center open-label single-arm study. The subjects will be enrolled and assigned into a single study group. Subjects will be required to complete four (4) treatment visits and four follow-up visits, 1 month, 3, 6 and 12 months after the final treatment.

At the baseline visit photographs of the abdomen will be taken. In addition, patient umbilical circumference will be measured and the subject's weight will be recorded. In addition, at the last therapy visit, subjects will receive Subject Satisfaction and Therapy Comfort Questionnaires to fill in.

Safety measures will include documentation of adverse events (AE) including subject's experience of pain or discomfort after the procedure. Following each treatment administration and at the follow-up visits, subjects will be checked for immediate post-procedure adverse event assessment.

Post-procedure evaluation (follow-up visits) will be conducted 1 month, 3, 6 and 12 months after the final treatment. Umbilical circumference and weight measure will be conducted at every follow-up visit. Also, subject's satisfaction will be noted. During the first (1 month), third (6 months) and last (12 months) follow-up visits, photographs of abdomen will be taken.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects of both genders with unwanted abdominal fat and expressing interest in treatment
* Age ≥ 22 years
* Voluntarily signed informed consent form
* BMI ≤ 30 kg/m2

Exclusion Criteria:

* Cardiac pacemakers
* Electronic implants
* Pulmonary insufficiency
* Metal implants
* Drug pumps
* Haemorrhagic conditions
* Anticoagulation therapy
* Heart disorders
* Malignant tumor
* Fever
* Pregnancy
* Breastfeeding
* Following recent surgical procedures when muscle contraction may disrupt the healing process
* Application over menstruating uterus
* Application over areas of the skin which lack normal sensation
* Scars, open lesions and wounds at the treatment area
* Unrepaired abdominal hernia

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2019-05-15 (Estimated); Study Completion 2019-06-15 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the device assessed through photography evaluation | 13 months
  Photography evaluations with correct identification of pre-treatment images compared to post-treatment images.
Effectiveness of the device assessed through change in adipose/muscle layer thickness | 13 months
  Change in umbilical circumference between pre-treatment and post-treatment based on waist circumference measure.
Subject's satisfaction | 13 months
  The 5-point Likert scale Subject Satisfaction Questionnaire will be used for an analysis of the subject's opinion of the therapy results. Subjects will be evaluating agreement with three different statements (concerning satisfaction with therapy results and appearance of abdominal area after therapy) by choosing an answer on a scale between 1 (Strongly disagree) and 5 (Strongly agree). Minimally 80% of the treated subjects should report the agreement with all three statements given in the questionnaire (answers "Agree" and "Strongly agree") in order to claim subject's satisfaction with the therapy outcome.

SECONDARY OUTCOMES:
Safety of the device for non-invasive fat disruption | 13 months
  The secondary objective of the study is to determine side effects and adverse events (AE) associated with the treatment of the abdominal area.
  The occurrence of adverse events will be followed throughout the whole study.
Therapy comfort | 3 months
  Therapy comfort will be noted at the last therapy visit. Subjects will be asked to evaluate the agreement with the statement concerning the conformity of the study treatment. Subjects will be evaluating the agreement by choosing an answer on a scale between 1 (Strongly disagree) and 5 (Strongly agree). Based on a given answers, the therapy comfort will be calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- Chicago Cosmetic Surgery and Dermatology, Chicago, Illinois, United States
- Derma Vita Clinic, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No